CLINICAL TRIAL: NCT07335614
Title: An Open Label, Single Center Study to Evaluate the Effect of Protein Loading on the Measurement of Renal Reserve Using the MediBeacon® Transdermal GFR System
Brief Title: Evaluation of Protein Loading on Measurement of Renal Reserve
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 100-301
Record Dates: First submitted 2025-12-23; First posted 2026-01-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Glomerular Filtration Rate
Keywords: Relmapirazin; Lumitrace

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 130 mg Lumitrace (Experimental): Participants will have the TGFR sensor placed and background measurements initiated. Participants will then receive a single intravenous 130 mg dose of Lumitrace. Approximately three hours later, they will ingest a high protein meal consisting of approximately 1.25 g/kg in a protein shake over 15-20 minutes following a minimum of an 8 hour fast. They will be followed at the study center for up to 6-8 hours following administration of Lumitrace.
  Interventions: Device: Lumitrace; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR)

INTERVENTIONS:
Device: Lumitrace — 18.6 mg/mL in a 7.0 mL volume administered by intravenous injection over 30 - 60 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 - 60 seconds
  Other Names: Relmapirazin
Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR) — Site staff will place and affix the TGFR reusable sensor and Disposable Ring for all enrolled participants. One sensor will be attached to the upper chest. An adhesive clip, surgical tape or other means may also be used to alleviate tension on the sensor cord. TGFR assessments will be collected for a minimum of 6 hours up to 8 hours post Lumitrace injection.

SUMMARY:
The goal of this clinical trial is to evaluate the effect of protein loading on the measurement of renal reserve using the MediBeacon Transdermal glomerular filtration rate (tGFR) system. Adults with estimated glomerular filtration rate (eGFR) >30 ml/min/1.73 m^2 will be recruited to join the study. This is a potential new use for the tGFR for the assessment of renal reserve. Renal reserve is the increase in GFR that occurs in response to various stimuli, such as when one kidney is removed. The remaining kidney will often show an increase in GFR to compensate. Renal reserve is typically measured after a high protein meal and requires a reproducible stimulus and a repeated measurement of GFR.

The main questions it aims to answer are:

* To characterize the effect of protein loading on GFR (dose response curve) as assessed by the MediBeacon Transdermal GFR System
* To determine Renal Reserve in participants with chronic kidney disease (CKD) using the MediBeacon Transdermal GFR System
* To demonstrate whether any change in GFR following the protein stimulus is associated with a change in cardiac output using non-invasive bioimpedance (NICaS)

Participants will participate in a Screening visit that will take place within 28 days of the scheduled administration of Lumitrace. On dosing day, participants will have the tGFR reusable sensor with disposable adhesive ring placed on their chest, and the MediBeacon Transdermal GFR System initiated to collect background fluorescence. Following an injection of Lumitrace and the initiation of GFR assessments, participants will ingest a high protein meal over 15-20 minutes. They will be followed at the study center for up to 6-8 hours following administration of Lumitrace. All participants will participate in a follow-up phone call approximately 7 days after the last exposure to Lumitrace. Researchers will analyze the results to see if there is a detectable difference in fluorescence clearance rate following the high protein meal.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry, all participants must satisfy all of the following criteria:

1. Age > 18 years - male or female

   1. Eligible female non-pregnant participants who are either not of child-bearing potential or willing to use adequate contraception during the trial
   2. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post-dose
   3. For women of child-bearing potential, the participant should have a negative pregnancy test, and agrees to one of the following acceptable contraceptive methods used consistently and correctly i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization
   4. Men will not donate sperm during the study and for 1 month following the last dose of study drug
2. Participants who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
3. eGFR >30 mL/min/1.73 m^2
4. Capable of fasting for at least 8 hours prior to the evaluation day

Exclusion Criteria:

1. Current use of renin-angiotensin-aldosterone system inhibitors (RAASi) including angiotensin-receptor blockers (ARBs), angiotensin-converting enzyme inhibitors (ACE-inhibitors) or direct renin inhibitors that can't be stopped at least 5 half-lives prior to the study day.
2. Current use of sodium-glucose cotransporter-2 (SGLT2) inhibitors such as bexaglifloxin, canagliflozin, dapagliflozin, empagliflozin, ertugliflozin or others that can't be stopped at least 5 half-lives prior to the study day.
3. Currently taking any drug classified as a sympathomimetic drug such as dobutamine, dopamine, norepinephrine, epinephrine, isoproterenol or others.
4. Current over the counter use of cold medications containing ephedrine or weight loss drugs containing ephedra alkaloids
5. Current history of drug use involving cocaine, mephedrone, amphetamines or methamphetamine
6. The participant has participated in a clinical trial and has received an investigational product within the following time ranges: prior to the first dosing day in the current study: either 30 days or 5 half-lives of the investigational product (whichever duration is longer).
7. History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
8. History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, Lumitrace or other related products (intolerance to a drug is not considered a drug allergy).
9. Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial.
10. Significant scarring, tattoos or alterations in pigmentation on the sternum or other sensor location testing areas that would alter sensor readings versus other areas of the skin
11. Use of tanning sprays, tanning products etc. on the upper chest within 2 weeks of dosing day
12. Use make-up, lotions, Vaseline or other products on the upper chest on the day prior to or the day of assessments
13. Any serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, or psychiatric condition that in the opinion of the investigator would limit the subjects' ability to complete study requirements or may put the subject at increased risk or compromise the interpretability of study results.
14. Participants with positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Renal reserve percentage | Day 1
  Renal reserve (%) will be calculated as Peak glomerular filtration rate (GFR) during the assessment period minus the average baseline GFR/average baseline GFR.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Dorshow, PhD, Study Director — MediBeacon, Inc.
Locations (1):
- Fletcher Allen Health Care, University of Vermont Medical School, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No